CLINICAL TRIAL: NCT04108585
Title: Investigation of the Efficacy of Different Respiratory Methods in the Treatment of Patients With Respiratory Failure
Brief Title: Efficacy of Different Respiratory Methods in Intensive Care
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Prof Mehmet Turan Inal, Member of Intensive Care, Trakya University
Other Study IDs: TUTF-BAEK 2016-197
Record Dates: First submitted 2019-09-03; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HFO group: HFO therapy
  Interventions: Procedure: HFO therapy
- CPAP group: CPAP therapy
  Interventions: Procedure: CPAP therapy

INTERVENTIONS:
Procedure: HFO therapy — HFO therapy from mechanical ventilation
  Groups: HFO group
Procedure: CPAP therapy — CPAP therapy from mechanical ventilation
  Groups: CPAP group

SUMMARY:
Peripheral oxygen saturation, non-invasive blood pressure, heart rate, respiratory rate and respiratory rate are routinely used in our intensive care unit in the follow-up of patients. In the study, the patient papers will be followed and the respiratory support of the patients will be recorded and all follow-ups will be made from the patient follow-up chart. The aim of this study is to compare the CPAP and HFO methods.

DETAILED DESCRIPTION:
Respiratory insufficiency is frequently present in patients who are admitted to intensive care units and respiratory support is provided through respiratory device. Respiratory support can be given by intubating the patient or without intubating the patient.

It is a procedure with intubation complications and stimulation of the sympathetic system as well as tongue, lip and tooth injuries. In recent years, non-invasive respiratory support can be given with the aid of a mask or nasal cannula without intubation, which has stable hemodynamics, no secretion, can cough, adhere to orders, no face, neck and head injuries (difficulty in mask application) and the use of this method is rapidly increasing in intensive care units.

Non-invasive respiratory support can be provided by CPAP method. In this method, positive pressure blended oxygen can be given to the patient by using an oranasal mask. In the literature, the use of non-invasive CPAP has been reported to be the gold standard for respiratory failure, particularly in COPD and immunosuppressed patients. CPAP method is available as standard in mechanical ventilators used in intensive care. The major disadvantage of CPAP is the discomfort caused by the mask attached to the patient's face.

In recent years, high-flow oxygen therapy (HFO) has been introduced, and in this mode, high-flow oxygen therapy is applied to the patient with high frequency nasal route and especially successful in COPD patients. In this method, patient comfort is higher since there is no mask attachment. The HFO device is not available in the intensive care unit and is planned to be purchased with the support of TUBAP.

In our intensive care unit, patients are primarily given non-invasive respiratory support. Follow-up during this support is extremely important. Whether the non-invasive respiratory support is sufficient is determined by follow-up. Following non-invasive respiratory support, patients are followed up, respiratory frequency rises above 30-35 in the first hour, peripheral oxygen saturation <90% decrease, systolic blood pressure increase 20%, 180 mmHg rise below 90 mmHg In case of an increase in heart rate of 20 beats / min, heart rate of more than 140 beats per minute, tachypnea, intercostal withdrawal, agitation and distress, the patient is intubated and respiratory support is applied invasively. Peripheral oxygen saturation, non-invasive blood pressure, heart rate, respiratory rate and respiratory rate are routinely used in our intensive care unit in the follow-up of patients. In the study, the patient papers will be followed and the respiratory support of the patients will be recorded and all follow-ups will be made from the patient follow-up chart. The aim of this study is to compare two different non-invasive breathing methods.

ELIGIBILITY:
Inclusion Criteria:

1. They have completed the age of 18
2. need oxygen therapy due to respiratory failure
3. Hemodynamic stability
4. Coughing
5. follow orders
6. face, neck and head without injury

Exclusion Criteria:

1. To be under 18 years
2. pregnant women
3. nursing

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  1. They have completed the age of 18
  2. need oxygen therapy due to respiratory failure
  3. Hemodynamic stability
  4. Coughing
  5. follow orders
  6. face, neck and head without injury
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Heart rate as per minute | Change from Baseline Heart rate as per minute at 1.hour
  variable 1
peripheral oxygen saturation as % value | Change from Baseline peripheral oxygen saturation as % value at 1.hour
  variable 2
arterial blood pressure as mmHg value | Change from Baseline arterial blood pressure as mmHg value at 1.hour
  variable 3

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brotfain E, Zlotnik A, Schwartz A, Frenkel A, Koyfman L, Gruenbaum SE, Klein M. Comparison of the effectiveness of high flow nasal oxygen cannula vs. standard non-rebreather oxygen face mask in post-extubation intensive care unit patients. Isr Med Assoc J. 2014 Nov;16(11):718-22. PMID 25558703